CLINICAL TRIAL: NCT02081989
Title: Effect of Renal Sympathetic Denervation on Glycemic Status Independent of Blood Pressure-lowering.
Brief Title: Renal Denervation in Diabetes.
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to commence study due to closure of hospital department.
Sponsor: Monash University (Other)
Collaborators: National Heart Foundation, Australia (Other)
Responsible Party: Principal Investigator, Ingrid Hopper, Senior Lecturer, Monash University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-01/13; 256/13 (Other: Alfred Hospital)
Record Dates: First submitted 2014-03-06; First posted 2014-03-07 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes
Keywords: Diabetes; Renal denervation
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Denervation (Experimental): Renal denervation
  Interventions: Procedure: Renal denervation
- No intervention (No Intervention): Control group - no intervention

INTERVENTIONS:
Procedure: Renal denervation — Renal denervation
  Arms: Denervation

SUMMARY:
Renal denervation (the use of radio waves to oblate the renal artery) has been shown to be an effective treatment for high blood pressure. It is currently being tested in heart failure patients and we would now like to look it its effects on diabetes.

We therefore plan to enrol 20 participants with type II diabetes into this study. Half will undergo renal denervation in addition to their standard care and the other half will act as controls and only receive standard care. Treatment allocation will be randomly assigned.

All participants will undergo screening (including a physical exam, blood tests, ultrasounds and a muscle biopsy). All patients will have follow up tests (including physical exams and blood tests) 1, 3 and 6 months later.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* Able and willing to provide informed consent
* Patients with established type II diabetes mellitus (HbA1C>7%, diet or oral hypoglycaemic agents)
* Clinical stable as demonstrated by no change in background anti-diabetic medication in the last 30 days.
* Anticipated that patients are able to maintain a stable dose of medication for the duration of the study

Exclusion Criteria:

* Renal arterial anatomy ineligible for RDN: main renal arteries <4 mm in diameter or <20 mm in treatable length; multiple renal arteries where main renal artery is estimated to supply <75% of the kidney; haemodynamically or anatomically significant renal artery abnormality or stenosis in either renal artery which, in the investigator's opinion, would interfere with safe cannulation of the renal artery or require surgical repair or interventional dilation
* History of prior renal artery intervention including balloon angioplasty, stenting or previous renal denervation.
* Single functioning kidney
* Need for insulin (interferes with euglycemic clamp testing) or GLP-I analogues
* eGFR <30 ml/min (MDRD formula)
* Any medical condition which, in the investigators opinion, may adversely affect the participants safety in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Glycemic control | 6 months
  Change in glycemic control at 6 months.
glucose uptake into peripheral skeletal muscle | 6 months
  To assess glucose uptake into peripheral skeletal muscle

CONTACTS AND LOCATIONS:
Overall Officials: Henry Krum, MBBS, FRACP, PhD, Principal Investigator — Monash University / Alfred Hospital
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia